CLINICAL TRIAL: NCT06655012
Title: The Muscle Anabolic Response to β2-adrenergic Stimulation
Brief Title: Salmeterol Effect on Exercise Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SALM_acute
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Beta2-adrenergic stimulation; Skeletal muscle hypertrophy
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Salmeterol (Experimental): Participants are administered salmeterol from an inhaler device
  Interventions: Drug: Salmeterol
- Placebo (Placebo Comparator): Participants are administered placebo from an inhaler device
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salmeterol — Participants are administered 200 µg salmeterol (8 puffs) from a MDI device
  Arms: Salmeterol
Drug: Placebo — Participants are administered placebo (8 puffs) from a MDI device
  Arms: Placebo

SUMMARY:
The purpose of the project is to investigate the muscle anabolic response to acute beta2-adrenergic stimulation in young healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* Age 18-40
* Physically active >5 hours a week
* Maximum oxygen uptake classified as high or very high

Exclusion Criteria:

* Active smoker currently or within the past 5 years
* Regular intake of medication deemed by the responsible study physician to affect the test parameters (hormonal contraception is accepted for women)
* Chronic or acute illness deemed by the responsible study physician to affect the test parameters
* Deviation from the study protocol
* Lean mass index >21 kg/m²
* Pregnancy
* Smoker
* Blood donation during the past 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Power output during sprint testing | Through study completion, an average on 2 weeks
  Power output measured in Watts during a sprint on a bike ergometer

SECONDARY OUTCOMES:
Power output during time trial | Through study completion, an average on 2 weeks
  Mean power output measured in Watts during a time trial on a bike ergometer

OTHER OUTCOMES:
Quadriceps strength | Through study completion, an average on 2 weeks
  Maksimal torque (Nm) achieved during isometric contraction

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided